CLINICAL TRIAL: NCT01709604
Title: The Efficacy and Safety of Continuous Venovenous Hemofiltration in Patients With Severe Acute Paraquat Poisoning
Brief Title: Role of CVVH in Patients With Acute Paraquat Poisoning
Acronym: PQ
Status: Completed | Type: Observational
Sponsor: Ai Peng (Other)
Responsible Party: Sponsor-Investigator, Ai Peng, Director of the department of Nephrology, Shanghai 10th poeple's hospital, Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Other Study IDs: 20120830; 8117192 (Other Grant/Funding Number: NSFC)
Record Dates: First submitted 2012-10-11; First posted 2012-10-18 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Poisoning by Paraquat With Undetermined Intent
Keywords: acute paraquat poisoning; hemoperfusion; continuous blood purification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Plasma, Urine,Dialysate
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- continuous venovenous hemofiltration: Continuous venovenous hemofiltration(CVVH):blood access was achieved by placing a double lumen catheter in the femoral or internal jugular vein. Continuous diffusive solute transport is achieved by infusing a dialysis fluid that runs counter-current to blood at an ultrafiltration rate of 35 ml/h/Kg.
  Interventions: Procedure: CVVH
- Standardized therapy regimens: The standardized therapy regimens included reduce absorption, accelerate the elimination and prevent the complications in patients with paraquat poisoning.
  Interventions: Procedure: CVVH; Procedure: Standardized therapy regimens

INTERVENTIONS:
Procedure: CVVH — Ultrafiltration at 35ml/h/Kg
  Other Names: continuous renal replacement treatment(CRRT); continuous blood purification(CBP)
Procedure: Standardized therapy regimens — Standardized therapy regimens included the followings:
  1. Remove all contaminated clothing
  2. Gastric lavage
  3. Receive activated charcoal as quickly as possible
  4. Hemoperfusion with activated charcoal(160g)
  5. Immunosuppression with methylprednisolone
  6. Antioxidants (glutathione,1.2 gram iv twice a day)
  7. Supportive care
  Groups: Standardized therapy regimens

SUMMARY:
Paraquat poisoning is characterized by multiple organ failure and pulmonary fibrosis with respiratory failure. Accumulating evidence suggested that continuous venovenous hemofiltration (CVVH) had a beneficial role in the treatment of multiple organ dysfunction. The investigators hypothesized that CVVH might restore multiple organ function and reduce the high mortality rate of paraquat poisoning. To confirm it, an prospective clinical study would be carried out.

DETAILED DESCRIPTION:
Paraquat (1,1 '-dimethyl-4,4'-bipyridylium dichloride) is widely used as a herbicide. Accidental or intentional ingestion of paraquat is common in many developing countries such as China, Sri Lanka and Korea because of easy access. The high mortality rate of paraquat is due to its high toxicity and the lack of effective treatments. Thus, the paraquat poisoning becomes one of major medical problem in the developing countries.

Paraquat poisoning is also one of major causes of death among young patients with acute poisoning in China. It is characterized by multiple organ failure and pulmonary fibrosis with respiratory failure. A growing body of evidence suggested that continuous venovenous hemofiltration (CVVH) had a great beneficial role in the treatment of multiple organ dysfunctions. We hypothesized that CVVH might reduce the high mortality rate of paraquat poisoning via restoring the multiorgan function, such as acute hepatic lesion, acute kidney injury, acute lung injury and acute pancreatic injury. We expect to enroll 100 patients from our hospital within 1 week after oral intake of paraquat. All patients were divided into Group 1 and Group 2. Group 1 were treated with a standardized therapeutic regimen including stomach lavage, emergency haemoperfusion and drugs. Group 2 were accepted with standardized treatment plus CVVH. The aim of this prospective clinical study was to evaluate the safety and efficacy of CVVH for the treatment of patients with paraquat poisoning. The survival rate, clinical manifestations and clinical parameters between these two groups were compared.

ELIGIBILITY:
Inclusion Criteria:

* All patients recruited in this study should meet the requirements as follows:

  1. history of exposure to Paraquat
  2. concentration in urine or plasma from all patients who arrived at our hospital within 1 week of paraquat ingestion was more than 0.1 mg/L.
  3. Patients with a light blue, navy blue or dark blue color in urine dithionite tests within 1 week of PQ ingestion, were classified as having PQ intoxication and were included in this study.
  4. patients with acute organ dysfunction such as acute kidney injury, hepatic injury or pancreatic injury.

     Exclusion Criteria:

Patients who had colorless urine PQ tests, who arrived at any hospital more than 24 h after intoxication, who had not orally ingested PQ or any other drug poisonings, who were younger than 14 years or older than 70 years, or who had been included in any previous control trials were excluded.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In-patients with acute paraquat poisoning
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2012-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Efficacy | at 6 months after paraquat poisoning
  CVVH treatment efficacy was assessed by the following measurements:
  1. Mortality rate: compared the difference between standardized therapy and CVVH treatment.
  2. Number of organs involved in paraquat poisoning such as lung,kidney,liver and heart.
  3. Degree of organ injuries
  4. CT scan of lung
  5. Biomarkers:
  1)Oxidative stress: blood superoxide dismutase(SOD),malondialdehyde (MDA), superoxide dismutase (SOD), and catalase (CAT).
  2)Proinflammatory factors: interleukins(IL-2,IL-6,IL-8 and IL-10) 3)Kidney function:serum cystatin C and estimated glomerular filtration rate (eGFR) and N-acetyl-β-(D)-glucosaminidase activity (NAG),kidney injury molecule-1 (KIM-1), Neutrophil gelatinase-associated lipocalin(NAGL) and urinary retinol-binding protein(RBP),etc.
  4)Heart damage markers: cTnT，MYO，creatine kinase-MB(CK-MB) and brain natriuretic peptide(BNP).

SECONDARY OUTCOMES:
Safety of CVVH for the treatment of patients | at 2 weeks after paraquat poisoning
  Safety and tolerability were assessed by the followings.
  1. Changes from baseline in systolic blood pressure and mean artery pressure during CVVH treatment procedure.
  2. Number of participants with adverse events such as bleeding, respiratory failure,hypotension,shock,thrombosis,pulmonary embolism and death.

CONTACTS AND LOCATIONS:
Overall Officials: Ai Peng, Ph.D., M.D., Principal Investigator — Shanghai 10th People's Hospital
Locations (2):
- China (2):
  - The division of nephrolgoy, Shanghai 10th people's hospital, Shanghai, Shanghai Municipality
  - The division of nephrology, Shanghai 10th people's hosptial, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No